CLINICAL TRIAL: NCT00597896
Title: Cognitive Enhancement in Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Ray, Susan, Senior Research Coordinator, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-069; 05T-670 (Other Grant/Funding Number: Stanley Medical Research Institute)
Record Dates: First submitted 2008-01-08; First posted 2008-01-18 (Estimated); Results first posted 2015-06-12 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Pramipexole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active pramipexole (Experimental): Day 1: Random assignment to drug or placebo and dosage starting at 0.125 mg BID, which will be increased every week to a target dose of 1.5 mg/day. Targeted maximum dose of 1.5 mg/day is expected to be reached by week 4, however, dosing will be flexible based upon side effects reported. The maximum dose will be 1.5 mg/day.
  Interventions: Drug: pramipexole
- Placebo pramipexole (Placebo Comparator): Day 1: Random assignment to drug or placebo and dosage starting at 0.125 mg BID, which will be increased every week to a target dose of 1.5 mg/day. Targeted maximum dose of 1.5 mg/day is expected to be reached by week 4, however, dosing will be flexible based upon side effects reported. The maximum dose will be 1.5 mg/day.
  Interventions: Drug: pramipexole

INTERVENTIONS:
Drug: pramipexole — po pramipexole versus matching placebo minimum 0.125 mg bid and maximum 0.75 mg bid
  Other Names: Mirapex

SUMMARY:
The purpose of this study is to examine whether the medication pramipexole (Mirapex) may be able to improve cognitive problems (i.e. difficulties with thinking, memory, and concentration) that may be associated with bipolar disorder.

DETAILED DESCRIPTION:
To address the primary aim, the study is an eight-week, randomized, double-blind, placebo-controlled treatment trial of pramipexole in 50 euthymic bipolar I and II disorder (BPD) patients, who demonstrate cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 18 and 65 years of age, who meet Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) criteria for BPD I or II (by SCID) and confirmed in the diagnostic consensus conference will be included.
* Subjects must also meet criteria for euthymia described above.
* All subjects must be taking a standard mood stabilizer at a stable therapeutic dose (i.e. lithium, carbamazepine, valproate, lamotrigine).

Exclusion Criteria:

* Subjects with a history of central nervous system (CNS) trauma, neurological disorder, Attention Deficit Hyperactivity Disorder (ADHD), or learning disability will be excluded.
* Subjects with a DSM-IV diagnosis of current or recent substance abuse or dependence (in the previous 1 month) will be excluded.
* Moreover, subjects with rapid-cycling during the past year will be excluded (based on SCID).
* Any subject with an active, unstable medical problem that may interfere with cognition will be excluded based on the investigator's judgment.
* While medication status is an important consideration in any study of bipolar disorder, the exclusion of patients taking any medication is not practical, given the high prevalence of combination pharmacotherapy for bipolar disorder. To help control for medication effects on cognition, we plan to limit the types of medications allowed by excluding certain medications with a known impact on cognitive performance.

  * Subjects taking clozapine will be excluded due to it's potential overlapping mechanisms of action with pramipexole.
  * Subjects taking prescription or over-the counter medications may also be excluded if these medications have been shown to impact cognition (i.e. diphenhydramine).
  * The use of benzodiazepines, sedatives, or sleeping pills, within 6 hours of neurocognitive testing will not be allowed. In addition, patients taking topiramate, tricyclic antidepressants, or anticholinergic medications that are known to impact cognition will be excluded from participation.
  * Subjects taking any medications that are known to interact with pramipexole (i.e. Zantac, Tagamet, Reglan, Benemid, Probalan, Compazine, Phenergan, quinidine, selegiline, verapamil, and any other medication with a known interaction) will also be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anil K. Malhotra, MD, Principal Investigator — Northwell Health; Katherine Burdick, PhD, Principal Investigator — Northwell Health
Locations (1):
- North Shore - Long Island Jewish Health System, Glen Oaks, New York, United States

REFERENCES:
- [Result] Burdick KE, Braga RJ, Nnadi CU, Shaya Y, Stearns WH, Malhotra AK. Placebo-controlled adjunctive trial of pramipexole in patients with bipolar disorder: targeting cognitive dysfunction. J Clin Psychiatry. 2012 Jan;73(1):103-12. doi: 10.4088/JCP.11m07299. Epub 2011 Nov 29. PMID 22152405

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Pramipexole: 0.125 mg BID-0.75 mg BID pramipexole
- Placebo Pramipexole: 0.125 mg BID-0.75 mg BID - matching placebo
Period: Overall Study
Arm/Group | Active Pramipexole | Placebo Pramipexole
Started | 24 | 26
Completed | 21 | 24
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Active Pramipexole: 0.125 mg BID-0.75 mg BID - pramipexole
- Total: Total of all reporting groups
Arm/Group | Active Pramipexole | Placebo Pramipexole | Total
Number analyzed (Participants) | 21 | 24 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 24 | 45
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.81 (9.4) | 44.42 (12.2) | 44.14 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 7 | 14 | 21
Region of Enrollment [Number; unit: participants]
  United States | 21 | 24 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in Weschler Adult Intelligence Scale-Third Edition (WAIS-III) Digit Span Subtest (Digits Forward)
Description: The examinee is read a sequence of numbers and must recall the numbers in the same order. Measures auditory attention and verbal working memory. The standard scores were reported for this measure. Values indicate the change from baseline to week 8, with positive values reflecting higher scores at week 8 and negative values reflecting lower scores at week 8.
Time Frame: Change from Baseline to Week 8
Population: All randomized participants were assessed per protocol
Measure: Mean (Standard Deviation); unit: number of correct numbers recalled
Arm/Group | Active Pramipexole | Placebo Pramipexole
Number analyzed (Participants) | 21 | 24
number of correct numbers recalled
  Baseline | 8.43 (2.93) | 8.54 (3.02)
  Week 8 | 8.48 (2.40) | 8.13 (2.52)
  Change from Baseline to Week 8 | .05 (1.72) | -.41 (2.08)

2. Secondary Outcome: Double-blind: Change From Baseline in Hamilton Rating Scale for Depression (HAM-D-21) Total Score at Endpoint
Description: The Hamilton Depression Rating Scale is a clinician-rated scale used to rate depression severity. The items are rated on either a 5-point (0 to 4) or a 3-point (0 to 2) scale. The 5-point scale uses a rating of 0 (absent), 1 (doubtful to mild), 2 (mild to moderate), 3 (moderate to severe), and 4 (very severe). Higher scores indicate worsening. The responses are summed to yield the HAM-D-21 score that ranges from 0-64.
Time Frame: Change from Baseline to Week 8
Population: All randomized participants were assessed per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Pramipexole | Placebo Pramipexole
Number analyzed (Participants) | 21 | 24
units on a scale | -.9 (5.5) | -1.5 (3.2)

3. Secondary Outcome: Double-blind: Change From Baseline in Clinician-Administered Rating Scale for Mania (CARS-M)Total Score at Endpoint
Description: The CARS-M is a 15-item clinician-rated scale designed to assess severity of both manic and psychotic symptoms. There are 2 subscales: a mania scale and a scale for psychotic symptoms and disorganization. There are a total of 15 items on the CARS-M, each of which is rated on a 6-point Likert scale (0/Absent to 5/Extreme), with the exception of item 15 ("Insight") which is rated on a 5-point Likert scale. These items yield two subscale scores-one for Mania (items 1-10) and one for Psychosis (items 11-15). Higher scores indicate worsening. The responses are summed to yield the CARS-M-15 score that ranges from 0-74.
Time Frame: Change from Baseline to Week 8
Population: All randomized participants were assessed per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Pramipexole | Placebo Pramipexole
Number analyzed (Participants) | 21 | 24
units on a scale | .5 (4.0) | -.9 (3.0)

4. Primary Outcome: Change From Baseline to Week 8 in Weschler Adult Intelligence Scale-Third Edition (WAIS-III) Digit Span Subtest (Digits Backward)
Description: The examinee is read a sequence of numbers and must recall the numbers in reverse order. Measures auditory attention and verbal working memory. The standard scores were reported for this measure. Values indicate the change from baseline to week 8, with positive values reflecting higher scores at week 8 and negative values reflecting lower scores at week 8.
Time Frame: Change from Baseline to Week 8
Population: All randomized participants were assessed per protocol
Measure: Mean (Standard Deviation); unit: number of correct numbers recalled
Arm/Group | Active Pramipexole | Placebo Pramipexole
Number analyzed (Participants) | 21 | 24
number of correct numbers recalled
  Baseline | 6.48 (2.09) | 6.46 (2.48)
  Week 8 | 6.86 (1.96) | 6.67 (3.09)
  Change from Baseline to Week 8 | .38 (2.33) | .21 (1.35)

5. Primary Outcome: Change From Baseline to Week 8 in Weschler Adult Intelligence Scale-Third Edition (WAIS-III) Digit Symbol Coding Test
Description: Using a key, the examinee copies symbols that are paired with numbers within a specified time limit. Measures visual scanning and graphomotor speed. The standard scores were reported for this measure. Values indicate the change from baseline to week 8, with positive values reflecting higher scores at week 8 and negative values reflecting lower scores at week 8.
Time Frame: Change from Baseline to Week 8
Population: All randomized participants were assessed per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Pramipexole | Placebo Pramipexole
Number analyzed (Participants) | 21 | 24
units on a scale
  Baseline | 8.52 (2.64) | 8.08 (2.83)
  Week 8 | 9.05 (3.46) | 8.75 (3.07)
  Change from Baseline to Week 8 | .52 (2.23) | .67 (1.86)

6. Primary Outcome: Change From Baseline to Week 8 in Stroop Color-Word Test
Description: The Stroop Color-Word Test consists of a word page with words printed in black ink, a color page with 'Xs' printed in color, and a color-word page where the color and the word do not match. The examinee reads the words or names the ink colors as quickly as possible within a time limit. Measures selective attention and inhibitory control. The raw scores (total number of words read) for each trial were reported for this measure. Values indicate the change from baseline to week 8, with positive values reflecting higher scores at week 8 and negative values reflecting lower scores at week 8.
Time Frame: Change from Baseline to Week 8
Population: All randomized participants were assessed per protocol
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Active Pramipexole | Placebo Pramipexole
Number analyzed (Participants) | 21 | 24
words
  Word-Baseline | 99.95 (18.20) | 95.42 (13.16)
  Word-Week 8 | 103.10 (16.09) | 94.33 (14.40)
  Word- Change from Baseline to Week 8 | 3.14 (12.46) | -1.08 (10.08)
  Color- Baseline | 68.10 (16.75) | 66.54 (12.56)
  Color-Week 8 | 72.24 (15.36) | 66.29 (12.87)
  Color- Change from Baseline to Week 8 | 4.14 (9.08) | -.25 (8.05)
  Color-Word- Baseline | 41.57 (9.93) | 39.29 (9.43)
  Color-Word-Week 8 | 43.95 (12.55) | 40.08 (10.14)
  Color-Word-Change from Baseline to Week 8 | 2.38 (8.96) | .79 (6.32)

7. Primary Outcome: Change From Baseline to Week 8 in Trail Making Test Part A
Description: The examinee is instructed to connect a set of 25 dots as quickly as possible while maintaining accuracy. Measures attentional resources and is a measure of the frontal lobe "executive" functions of visual search, set-switching and conceptual flexibility. The total time in seconds was reported for this measure. Values indicate the change from baseline to week 8, with positive values reflecting higher scores at week 8 and negative values reflecting lower scores at week 8.
Time Frame: Change from Baseline to Week 8
Population: All randomized participants were assessed per protocol
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Active Pramipexole | Placebo Pramipexole
Number analyzed (Participants) | 21 | 24
seconds
  Baseline | 32.88 (15.66) | 35.37 (12.36)
  Week 8 | 28.57 (12.05) | 32.79 (13.99)
  Change from Baseline to Week 8 | -4.31 (8.23) | -2.58 (13.48)

8. Primary Outcome: Change From Baseline to Week 8 in Trail Making Test Part B
Description: The examinee is instructed to connect a set of 25 dots, alternating between numbers and letters, as quickly as possible while maintaining accuracy. Measures attentional resources and is a measure of the frontal lobe "executive" functions of visual search, set-switching and conceptual flexibility. The total time in seconds was reported for this measure. Values indicate the change from baseline to week 8, with positive values reflecting higher scores at week 8 and negative values reflecting lower scores at week 8.
Time Frame: Change from Baseline to Week 8
Population: All randomized participants were assessed per protocol
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Active Pramipexole | Placebo Pramipexole
Number analyzed (Participants) | 21 | 24
seconds
  Baseline | 76.90 (30.64) | 106.14 (75.30)
  Week 8 | 75.55 (34.52) | 93.39 (73.09)
  Change from Baseline to Week 8 | -1.35 (28.48) | -12.74 (43.76)

9. Primary Outcome: Change From Baseline to Week 8 in d2 Test of Attention
Description: The d2 Test of Attention consist of 14 lines, each comprised of 47 characters, for a total of 658 items. The examinee must scan each line and cross out all the "d's" with two dashes. The subject is allowed 20 seconds per line. Measures rapid processing of visual information and motor speed.
Time Frame: Change from Baseline to Week 8
Population: All randomized participants were assessed per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Pramipexole | Placebo Pramipexole
Number analyzed (Participants) | 21 | 24
units on a scale | .90 (6.84) | 1.54 (7.91)

10. Primary Outcome: Change From Baseline to Week 8 in Hopkins Verbal Learning Test
Description: The examinee is required to recall a list of 12 words over 3 immediate learning trials, a delayed recall trial and a recognition trial. Measures learning and retention of verbal material. The total number of words recalled during the delayed recall trial was reported. Values indicate the change from baseline to week 8, with positive values reflecting higher scores at week 8 and negative values reflecting lower scores at week 8.
Time Frame: Change from Baseline to Week 8
Population: All randomized participants were assessed per protocol
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Active Pramipexole | Placebo Pramipexole
Number analyzed (Participants) | 21 | 24
words
  Baseline | 8.00 (2.17) | 8.13 (2.61)
  Week 8 | 8.09 (2.86) | 8.42 (2.34)
  Change from Baseline to Week 8 | .09 (2.55) | .29 (2.07)

11. Primary Outcome: Change From Baseline to Week 8 in Controlled Oral Word Association Test (COWAT) Letter Fluency
Description: The examinee is required to say as many words as they can think of in one minute that begin with a given letter of the alphabet. The task contains three trials. Measures phonetic verbal fluency. The raw score (total words recorded across the three trials) was reported. Values indicate the change from baseline to week 8, with positive values reflecting higher scores at week 8 and negative values reflecting lower scores at week 8.
Time Frame: Change from Baseline to Week 8
Population: All randomized participants were assessed per protocol
Measure: Mean (Standard Deviation); unit: words
Arm/Group | Active Pramipexole | Placebo Pramipexole
Number analyzed (Participants) | 21 | 24
words
  Baseline | 38.33 (13.48) | 33.63 (12.13)
  Week 8 | 39.62 (14.30) | 33.50 (10.49)
  Change from Baseline to Week 8 | 1.29 (6.76) | -.13 (8.74)

ADVERSE EVENTS:
Arm/Group | Active Pramipexole | Placebo Pramipexole
Serious Adverse Events (participants affected / at risk) | 2/21 | 1/24
Other Adverse Events (participants affected / at risk) | 0/21 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Pramipexole (N=21) | Placebo Pramipexole (N=24)
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Car accident (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes